CLINICAL TRIAL: NCT04792372
Title: Evaluation of the Effects of Initial Macrophage and Th17 Cell Activities on the Healing Following Periodontal Phase I Therapy
Brief Title: Evaluation of the Effects of Immune Cells on Periodontal Healing
Acronym: EMTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other); University of Turku (Other)
Responsible Party: Principal Investigator, Mustafa YILMAZ, Asst Prof, Biruni University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: TheMacPer
Record Dates: First submitted 2021-02-23; First posted 2021-03-11 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Periodontitis
Keywords: Periodontitis; Macrophages; T-Lymphocytes; Treatment Outcome
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Healing will be monitored of periodontitis patients who receive conventional initial treatment. The patients will be grouped according to their healing capacity at the end of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Periodontitis patients (Other): Single-group receiving periodontal treatment. The data will be evaluated according to the healing potential of individuals in the group and also site-specifically.
  Interventions: Procedure: Initial periodontal treatment

INTERVENTIONS:
Procedure: Initial periodontal treatment — Conventional periodontal treatment (scaling and root debridement) will be conducted

SUMMARY:
Periodontitis is an inflammatory disease with an infectious character, where, as the result of the host response to a dysbiotic microflora, attachment and bone loss occur. The host response and the healing period following the treatment differs among individuals, but the reason behind is not fully understood. The macrophages and T cells play an important role in the immune response and in the pathogenesis of periodontal diseases, but their role in the healing following periodontal therapy is not known. In this study, we aim to reveal the effects of initial macrophage and T cell activities in the gingival tissue on the differences of the response to phase I periodontal treatment.

42 individuals will be included in the study. Granulation tissue samples will be collected from two separate deep pockets of each individual, initially. At the same session, full-mouth scaling and root debridement will be conducted. Saliva, subgingival biofilm and gingival crevicular fluid (GCF) samples will also be collected, initially, and at the 2nd, 6th, 12th and 24th weeks. At the same appointments, periodontal parameters will be recorded. When the clinical procedures are concluded, the samples will be sent to Turku University with dry ice. Tissue and GCF concentrations of related cytokines will be analyzed with Luminex. The density of macrophage types will be defined by immunoblot analysis of related markers. Macrophage subpopulations in tissues will be specified by proteomics. Likewise, quantities of periodontal pathogens will be evaluated with DNA isolation and next generation sequencing.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe periodontitis
* having at least two pockets ≥ 6 mm
* systemic healthy

Exclusion Criteria:

* received periodontal treatment prior to study
* received antibiotic or antiinflammatory drugs in the last 6 months
* pregnant or in lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Probable pocket depth (PPD) | baseline, 2nd, 6th, 12th and 24th weeks following therapy
  distance between the gingival margin and pocket base (mm); full-mouth scores, 6 sites per tooth
Change in Bleeding on probing (BoP) | baseline, 2nd, 6th, 12th and 24th weeks following therapy
  visual inspection, dichotomous; full-mouth, 6 sites per tooth; change in positive sites %
Baseline macrophage related cytokine concentrations in granulation tissue samples | Samples will be obtained during the intervention and will be kept in -80oC until immunohistochemical analysis which will be carried out through study completion, 6-9 months
  two pockets (≥6mm; BoP+) of each individual; Luminex: monocyte chemoattractant protein (MCP)-1, -2, -3, -4; macrophage derived chemokine (MDC); macrophage inhibitory factor (MIF), monokine induced by gamma interferon (MIG), macrophage inflammatory protein (MIP)-1α, interferon γ-induced protein (IP)-10, CD163, TWEAK, BAFF concentrations (pg/mL); each will be correlated with the change in probable pocket depth and bleeding on probing scores
Baseline Th17-pathway related cytokine concentrations in granulation tissue samples | Samples will be obtained during the intervention and will be kept in -80oC until immunohistochemical analysis which will be carried out through study completion, 6-9 months
  two pockets (≥6mm; BoP+) of each individual; Luminex: Interleukin (IL)-1β, -4, -6, -10, -17A, -17F, -21, -22, -23, -25, -31, -33, interferon (IFN)-γ, soluble cluster of differentiation 40 ligand (sCD-40L), tumor necrosis factor (TNF)-ɑ concentrations (pg/mL); each will be correlated with the change in probable pocket depth and bleeding on probing scores
Baseline density of macrophage types in granulation tissue samples | Samples will be obtained during the intervention and will be kept in -80oC until immunohistochemical analysis which will be carried out through study completion, 6-9 months
  two pockets (≥6mm; BoP+) from each individual; Immunoblot analysis: cluster of differentiation(CD)68 and CD163; cell number / optic field (cells/mm2); each will be correlated with the change in probable pocket depth and bleeding on probing scores

SECONDARY OUTCOMES:
Change in macrophage and Th17-pathway related cytokine concentrations in saliva | baseline, 2nd, 6th, 12th and 24th weeks following therapy; immunohistochemical analysis will be carried out through study completion, 6-9 months
  MCP-1, -2, -3, -4, MDC, MIF, MIG, MIP-1α, IP-10, IL1β, -4, -6, -10, -17A, -17F, -21, -22, -23, -25, -31, -33, IFN-γ, sCD-40L, TNF-ɑ, sCD163, TWEAK, BAFF, sST2 concentrations (pg/mL); will be correlated with the change in probable pocket depth and bleeding on probing scores
Change in macrophage and Th17-pathway related cytokine concentrations in gingival crevicular fluid (GCF) | baseline, 2nd, 6th, 12th and 24th weeks following therapy; immunohistochemical analysis will be carried out when through study completion, 6-9 months
  MCP-1, -2, -3, -4, MDC, MIF, MIG, MIP-1α, IP-10, IL1β, -4, -6, -10, -17A, -17F, -21, -22, -23, -25, -31, -33, IFN-γ, sCD-40L, TNF-ɑ, sCD163, TWEAK, BAFF, sST2 concentrations (pg/mL); will be correlated with the change in probable pocket depth and bleeding on probing scores
Change in plaque index | baseline, 2nd, 6th, 12th and 24th weeks following therapy
  Silness-Löe plaque index (scored as 0-3); full-mouth, 6 sites per tooth; will be monitored for oral health assessment during the healing period
Change in clinical attachment level (CAL) | baseline, 2nd, 6th, 12th and 24th weeks following therapy
  distance between the cement-enamel junction and pocket base (mm); full-mouth, 6 sites per tooth; will be correlated with pocket depth reduction
Change in biofilm microbiota | baseline, 2nd, 6th, 12th and 24th weeks following therapy; microbiological analysis will be carried out through clinical phase completion, 6-9 months
  DNA isolation and next generation sequencing: P. gingivalis, T. denticola, T. forsythia, P. intermedia, F. nucleatum and A. actinomycetemcomitans; bacterial count (log10 scale)
Change in neutrophil-associated cytokines in saliva | baseline, 6th, 12th and 24th weeks following therapy
  MMP-2, MMP-7, MMP-8, active MMP-8, MMP-9, MMP-13, TIMP, myeloperoxidase, PMN elastase (IFMA and ELISA methods) concentrations (pg/mL) in saliva
Change in neutrophil-associated cytokines in and oral rinse | baseline, 6th, 12th and 24th weeks following therapy
  MMP-2, MMP-7, MMP-8, active MMP-8, MMP-9, MMP-13, TIMP, myeloperoxidase, PMN elastase (IFMA and ELISA methods) concentrations (pg/mL) in oral rinse samples
active MMP-8 point-of-care test results in oral rinse | baseline, 6th, 12th and 24th weeks following therapy
  Dichotomous aMMP-8 test results in oral rinse samples (according to the manufacturer, a concentration below 20 ng/mL gives a negative test result, otherwise positive - Periosafe (R) Dentognostics GmHb, Jena, Germany)

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa YILMAZ, Principal Investigator — Biruni University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No